CLINICAL TRIAL: NCT05187494
Title: A Study of the Role of Some Drug Delivery Systems in Enhancing the Efficiency of EMLA Cream in Palatal Anesthesia for Children Aged Between 7-11 Years Old
Brief Title: Enhancing the Efficiency of EMLA Cream in Palatal Anesthesia for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Pedo-05-2021
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Extrusion of Tooth
Keywords: EMLA; Micro-needle patches; Permeability enhancer; Oral patches
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Conventional local palatine injection (Other): Conventional palatal injection with anesthetic (lidocaine 2% with Epinephrine 1:80000, Korea) will be performed and the following measures (face expressions ( Wong-Baker Faces) heart rate and oxygen rate and FLACC pain scale) will be recorded to determine the reaction of the child.
  Interventions: Other: Conventional local palatine injection
- EMLA cream only (Experimental): The palatine mucosa will be dried with a cotton ball 2*2 and then 0,2 g of Emla cream will be applied for 3 minutes . During this period and the following measures (face expressions ( Wong-Baker Faces) heart rate and oxygen rate and FLACC pain scale) will be recorded to determine the reaction of the child.
  Interventions: Drug: EMLA cream only
- chemical permeability enhancer DMSO with EMLA cream (Experimental): The palatine mucosa will be dried with a cotton ball and then EMLA cream will be mixed with a permeability enhancer in the laboratory of pharmaceutical industries at the Faculty of Pharmacy at Damascus University according to the following: Adding 10 g of EMLA cream 5%, 1,026 g of DMSO 100% and it will be applied with cotton bud for a period of 3 minutes. During this period and the following measures (face expressions ( Wong-Baker Faces) heart rate and oxygen rate and FLACC pain scale) will be recorded to determine the reaction of the child.
  Interventions: Drug: chemical permeability enhancer DMSO with EMLA cream
- Oral patches with EMLA Cream (Experimental): The palatine mucosa will be dried with a cotton ball and then 0.2 g of EMLA cream 5% will be applied by using an oral patch 14*14 mm for 3 minutes. During this period and the following measures (face expressions ( Wong-Baker Faces) heart rate and oxygen rate and FLACC pain scale) will be recorded to determine the reaction of the child.
  Interventions: Drug: Oral patches with EMLA Cream
- Micro-needle patches dissolved with EMLA Cream (Experimental): The palatine mucosa will be dried with a cotton ball 2*2 and then 0.2 g of EMLA cream 5% will be applied by using an micro-needle patch 14*14 mm, 0,25 micron for 3 minutes.
  Interventions: Drug: Micro-needle patches dissolved with EMLA Cream

INTERVENTIONS:
Other: Conventional local palatine injection — Conventional palatal injection with anesthetic (lidocaine HCL2% with Epinephrine 1:80000, Korea) Then the palatal probe will be performed with a dental probe in contact with the bone to estimate anesthetic effectiveness
  Arms: Conventional local palatine injection
Drug: EMLA cream only — Emla cream will be applied at a distance of 1 mm from the palatine gingival edge by cotton buds for 3 minutes within the application area 14*14 mm and the mouth will be open throughout the procedure and the saliva will be controlled by a saliva absorbent. Then the palatal probe will be performed with a dental probe in contact with the bone to estimate anesthetic effectiveness.
  Arms: EMLA cream only
Drug: chemical permeability enhancer DMSO with EMLA cream — Adding 10 g of EMLA cream 5%, 1,026 g of DMSO 100% and it will be applied with cotton bud for a period of 3 minutes while the child is opening his mouth and the saliva is controlled by saliva absorbent. Then the palatal probe will be performed with a dental probe in contact with the bone to estimate anesthetic effectiveness.
  Arms: chemical permeability enhancer DMSO with EMLA cream
Drug: Oral patches with EMLA Cream — EMLA cream 5% will be applied at a distance of 1 mm from the palatal gingival edge using an oral patch 14*14 mm for 3 minutes and the Mouth will be closed throughout the procedure. Then the palatal probe will be performed with a dental probe in contact with the bone to estimate anesthetic effectiveness
  Arms: Oral patches with EMLA Cream
Drug: Micro-needle patches dissolved with EMLA Cream — EMLA cream 5% will be applied at a distance of 1 mm from the palatal gingival edge using an micro-needle patch 14*14 mm, 0,25 micron for 3 minutes and the Mouth will be closed throughout the procedure. Then the palatal probe will be performed with a dental probe in contact with the bone to estimate anesthetic effectiveness.
  Arms: Micro-needle patches dissolved with EMLA Cream

SUMMARY:
The aim of this study is to Avoid traditional palatal local injections when extracting upper primary teeth through enhancing the efficiency of EMLA cream by using drug delivery systems (permeability enhancer (DMSO), oral patches and micro-needle patches) for palatine injection.

Group 1: Conventional local palatine injection (control group). Group 2: EMLA cream only. Group 3 :chemical permeability enhancer DMSO with EMLA cream. Group 4: Oral patches with EMLA Cream. Group 5: Micro-needle patches dissolved with EMLA Cream.

DETAILED DESCRIPTION:
The insertion of the needle and the infusion of the anesthetic solution into the palate often uncomfortable for the children and their acceptance of dental treatment. Therefore, there is a need for studies to find ways to replace the palatine injection in the modern dentistry.

Effectiveness of Compound surfactant drugs (EMLA) have strong activity on the palatine tissues. Therefore, it will be chosen as an alternative to the traditional ones and will be enhanced by one of the drug delivery systems (physical/chemical).

Decreased permeability of the palatine mucosa is a major reason behind using drug delivery systems to reach an effective therapeutic level.

To our knowledge, this research will be the first which will be used a method of drug delivery systems to replace traditional palatal needle.

ELIGIBILITY:
Inclusion Criteria:

* no previous dental experience.
* Healthy children.
* Definitely positive or positive ratings of Frank scale
* Child did not receive any sedative or pain drugs during the last three.
* Presence of upper primary teeth, an indication for extraction

Exclusion Criteria:

* Presence of general diseases or health problems.
* Uncooperative children
* Children with congenital or idiopathic Methemoglobin
* Teeth with severe abscesses

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in the values of each of the heart rate and oxygen rate | On application of the substance
  The heart and oxygen rate will be recorded by pulse oximeter
Evaluation conventional local palatine injection | On palatal probing
  The heart and oxygen rate will be recorded by pulse oximeter
Evaluation conventional local palatine injection | On extraction
  The heart and oxygen rate will be recorded by pulse oximeter
Pain levels using self-reported Wong-Baker faces pain scale | On application of the substance
  0= "no hurt", 2= "hurts a little bit", 4="hurts a little more", 6= "hurts even more", 8= "hurts a whole lot", 10= "hurts worst"
Pain levels using self-reported Wong-Baker faces pain scale | On palatal probing
  0= "no hurt", 2= "hurts a little bit", 4="hurts a little more", 6= "hurts even more", 8= "hurts a whole lot", 10= "hurts worst"
Pain levels using self-reported Wong-Baker faces pain scale | On extraction
  0= "no hurt", 2= "hurts a little bit", 4="hurts a little more", 6= "hurts even more", 8= "hurts a whole lot", 10= "hurts worst"
Pain levels using FLACC scale | On application of the substance
  0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 =Moderate pain, 7-10 = Severe discomfort/pain
Pain levels using FLACC scale | On palatal probing
  0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 =Moderate pain, 7-10 = Severe discomfort/pain
Pain levels using FLACC scale | On extraction
  0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 =Moderate pain, 7-10 = Severe discomfort/pain

CONTACTS AND LOCATIONS:
Overall Officials: Farah M Babakurd, DDS, Principal Investigator — MSc student in Pedodontics, University of Damascus; Shadi K Azzawi, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munshi AK, Hegde AM, Latha R. Use of EMLA: is it an injection free alternative? J Clin Pediatr Dent. 2001 Spring;25(3):215-9. doi: 10.17796/jcpd.25.3.hn62713500418728. PMID 12049081
- [Background] Davidovich E, Wated A, Shapira J, Ram D. The influence of location of local anesthesia and complexity/duration of restorative treatment on children's behavior during dental treatment. Pediatr Dent. 2013 Jul-Aug;35(4):333-6. PMID 23930632
- [Background] Barcohana N, Duperon DF, Yashar M. The relationship of application time to EMLA efficacy. J Dent Child (Chic). 2003 Jan-Apr;70(1):51-4. PMID 12762609
- [Background] Franz-Montan M, Ribeiro LNM, Volpato MC, Cereda CMS, Groppo FC, Tofoli GR, de Araujo DR, Santi P, Padula C, de Paula E. Recent advances and perspectives in topical oral anesthesia. Expert Opin Drug Deliv. 2017 May;14(5):673-684. doi: 10.1080/17425247.2016.1227784. Epub 2016 Sep 1. PMID 27554455
- [Background] Shaikh R, Raj Singh TR, Garland MJ, Woolfson AD, Donnelly RF. Mucoadhesive drug delivery systems. J Pharm Bioallied Sci. 2011 Jan;3(1):89-100. doi: 10.4103/0975-7406.76478. PMID 21430958